CLINICAL TRIAL: NCT06814704
Title: Effect of Intraabdominal Hypopressive Exercises on Postnatal Backache and Functional Disability
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Salwa A. Shawat, Principle Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypopressive Exercises
Record Dates: First submitted 2024-02-14; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
Keywords: postpartum; low back pain; Quality of life
MeSH Terms: conditions — Low Back Pain | interventions — Acetaminophen; Diathermy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Experimental): Group A will receive 1. hypopressive abdominal exercises 2. traditional treatment for low back pain (Pharmacological treatment (paracetamol 0.5-1g 3times/day),Heat therapy Continuous low-level heat wrap(electrical) 3. Progressive strength training.
  Interventions: Other: Hypopressive exercises , hot packs, acetaminophen, progressive strengthening exercises
- Group (B) (Placebo Comparator): Group B will receive 1. traditional treatment for low back pain (Pharmacological treatment (paracetamol 0.5-1g 3times/day),Heat therapy Continuous low-level heat wrap(electrical) 2. Progressive strength training.
  Interventions: Other: heat therapy, pharmacological therapy, progressive strengthening exercises

INTERVENTIONS:
Other: Hypopressive exercises , hot packs, acetaminophen, progressive strengthening exercises — 20 subjects combined HE with traditional treatments for low back pain (heat therapy, medication, and progressive strength training).
  Arms: Group (A)
Other: heat therapy, pharmacological therapy, progressive strengthening exercises — Hypopressive exercises :The women were instructed to hold breath with chest extension for approximately 10 seconds before they began to breathe again. Then, using a series of upper and lower limb positions, the subjects were shown how to apply a series of "hypopressive postures
  Arms: Group (B)

SUMMARY:
The purpose of this study was to evaluate the effectiveness of hypopressive exercise in postpartum females with abnormal hyperlordosis and back pain.

Hypopressive exercises are safe and beneficial for new moms, as they can be started soon after delivery. They help strengthen postural muscles, reduce back pain, and manage pain by reducing intra-abdominal pressure, increasing activity of postural musculature, and normalizing myofascial tension.

DETAILED DESCRIPTION:
38 postpartum women with abnormal hyperlordosis. The women were then divided into two equal groups. Group A(n=19) received hypopressive abdominal exercise along with traditional treatment for lower back pain (LBP), while Group B(n=19) received the same treatment without hypopressive exercise. The main outcomes measured were the the Revised Short McGill Pain Questionnaire Version-2, the lumbar lordotic angle, and the patient-specific functional scale.

ELIGIBILITY:
Inclusion Criteria:

- participants must have a healthy pregnancy, a typical vaginal birth, LBP that existed 24 weeks after giving birth, and functional limitations in daily activities. The study only allowed women aged 20-35 with no more than two prior pregnancies and a BMI of less than 25 kg/m2 to participate.

Exclusion Criteria:

* women who under pharmacological or psychological treatment, had pelvic tumors, lumbar disk herniation, heart disease, hypertension, lumbar spine tumors, chronic uterine prolapse, chronic pelvic pain, lumbar spondylosis, or lumbar spondylolisthesis.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Pain assessment at the end of the study up to 8 weeks
  pain: The Revised Short McGill Pain Questionnaire will be used to assess both groups before and after the study.

SECONDARY OUTCOMES:
Assessment of functional disability | This scale will be done for each case at the end of the study up to 8 weeks
  The Patient-Specific Functional Scale (PSFS) will be used to assess functional changes in patients with musculoskeletal illnesses using self-reported data. Patients rated to five activities on an 11-point scale based on their current level of difficulty.

OTHER OUTCOMES:
Assessment of lumbar lordotic angle | It will be done for each case at the end of the study up to 8 weeks
  The angle will be measured using flexible ruler once before and once after the study by the primary examiner, who repeated each measurement three times.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh university, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
it need to have a permission from the faculty and university first